CLINICAL TRIAL: NCT00516243
Title: Phase IB Randomized, Double-Blinded, Placebo-Controlled, Dose Escalation Study of Polyphenon E in Women With a History of Hormone Receptor-Negative Breast Cancer
Brief Title: Defined Green Tea Catechin Extract in Treating Women With Hormone Receptor Negative Stage I-III Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00858; NCI-2009-00858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-AAAB7638; CDR0000653465; 2006-0521 (Other: M D Anderson Cancer Center); MDA04-4-01 (Other: DCP); P30CA016672 (NIH); N01CN35159 (NIH)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-04

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (defined green tea catechin extract) (Experimental): Patients receive defined green tea catechin extract PO BID for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: quality-of-life assessment; Procedure: questionnaire administration; Procedure: laboratory biomarker analysis; Drug: defined green tea catechin extract
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: quality-of-life assessment; Procedure: questionnaire administration; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: questionnaire administration — Ancillary studies
Procedure: laboratory biomarker analysis — Correlative studies
Drug: defined green tea catechin extract — Given PO
  Other Names: Polyphenon E
  Arms: Arm I (defined green tea catechin extract)

SUMMARY:
This randomized phase I trial studies the side effects and best dose of defined green tea catechin extract in treating women with hormone receptor-negative stage I-III breast cancer. Green tea extract contains ingredients that may prevent or slow the growth of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate the safety of green tea catechin extract (Polyphenon E) in women with a history of hormone receptor-negative breast cancer.

II. Determine the maximum tolerated dose of Polyphenon E in women with a history of hormone receptor-negative breast cancer.

SECONDARY OBJECTIVES:

I. Determine the efficacy of Polyphenon E in modulating histologic changes (nonproliferative, proliferative without atypia, atypical hyperplasia) on core biopsy of the contralateral breast.

II. Determine the efficacy of Polyphenon E in modulating immunohistochemical expression of Ki-67 (proliferation index), p53, EGFR, HER2/neu, cleaved caspase-3 (apoptosis marker), and estrogen receptor on core biopsy tissue of the contralateral breast.

III. Determine the efficacy of Polyphenon E in modulating mammographic breast density of the contralateral breast.

IV. Determine the efficacy of Polyphenon E in modulating hormone metabolites (serum estradiol, testosterone, IGF-1, IGFBP-3, SHBG).

V. Determine the efficacy of Polyphenon E in modulating eicosanoid levels (urine PGE-M).

VI. Determine the efficacy of Polyphenon E in modulating biomarkers of oxidative damage (urine 8-OHdG, isoprostane).

VII. Determine the efficacy of Polyphenon E in modulating serum C-reactive protein.

VIII. Determine the activity of Polyphenon E in relation to COMT genotype. IX. Assess quality of life and attitudes toward complementary and alternative medicine in women with a history of breast cancer.

OUTLINE: This is a dose-escalation study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive defined green tea catechin extract orally (PO) twice daily (BID) for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO BID for 6 months in the absence of disease progression or unacceptable toxicity.

Patients undergo a core biopsy and mammogram of the contralateral breast at baseline and after 6 months for histological evaluation, IHC analysis, and mammographic density reading. Core biopsy tissue is assessed for proliferative changes and presence of atypia using standardized histological criteria. Core biopsy tissue is also analyzed by IHC for the following proteins: Ki-67 (proliferation index), p53, EGFR, HER2/neu, cleaved caspase-3 (apoptosis marker), and estrogen receptor (ER). Blood and urine samples are collected at baseline and every 2 months during treatment to measure drug effect biomarkers: serum estradiol, testosterone, insulin-like growth factor-1 (IGF-1), IGF binding protein-3 (IGFBP-3), and sex hormone-binding globulin (SHBG) by immunological laboratory methods; urine prostaglandin levels (PGE-M) by tandem mass spectrometry; urine oxidative damage markers (8-OHdG, isoprostane) and serum C-reactive protein (CRP) by ELISA; and catechol-O-methyltransferase (COMT) genotype (at baseline only).

Patients complete a questionnaire assessing quality of life (SF-36) and attitudes toward complementary and alternative medicine at baseline and at 6 months.

After completion of study treatment, patients are followed for 1 month.

ELIGIBILITY:
Criteria:

* History of histologically confirmed stage I, II, or III breast carcinoma without evidence of disease at study entry
* No evidence of recurrent disease (patients with resected local recurrence are eligible)
* Normal mammogram of the contralateral breast within the past 12 months, defined as no new suspicious calcifications or other abnormal findings warranting a breast biopsy
* No history of histologically confirmed bilateral breast cancer
* No evidence of metastatic breast cancer
* Registered in the outpatient medical oncology clinic at Columbia University Medical Center (CUMC), MD Anderson Cancer Center (MDACC), Memorial Sloan Kettering Cancer Center (MSKCC), or the Weill-Cornell campus of New York Presbyterian Hospital (NYP-WC)
* Hormone receptor status: Estrogen- and progesterone-receptor negative
* Menopausal status: Pre- or postmenopausal
* ECOG performance status < 2 (Karnofsky > 60%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST/ALT =< 2.5 times institutional upper limit of normal
* Serum creatinine within normal institutional limits
* Not pregnant or nursing
* Negative pregnancy test
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to green tea extract (Polyphenon E), such as green tea food products or supplements containing EGCG
* No history of gastrointestinal bleeding including, but not limited to, any of the following: Diverticulosis; Peptic ulcer disease; Erosive gastritis; Varices
* No uncontrolled or significant co-morbid illness including, but not limited to, any of the following: active or serious infection requiring intravenous antibiotics; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; active gastrointestinal bleeding; active liver disease; psychiatric illness/social situations that would limit compliance with study requirements
* No active malignancy, except for squamous cell carcinoma of the skin; basal cell carcinoma of the skin; carcinoma in situ; stage IA or IB invasive squamous cell carcinoma of the cervix treated by surgery and/or radiation therapy; or stage IA grade 1 adenocarcinoma of the endometrium treated by surgery
* At least 6 months since prior chemotherapy, radiation therapy, and/or breast surgery
* No prior radiation therapy or implant in the contralateral breast
* More than 30 days since prior and no concurrent medications, herbs, or vitamin and mineral supplements that contain tea compounds or caffeine
* At least 30 days since prior and no other concurrent investigational agents
* At least 30 days since prior and no concurrent tea consumption
* Willing to limit regular coffee consumption to =< three 8-ounce cups per day for 30 days prior to baseline evaluation and during the study intervention
* Total daily caffeine consumption should not exceed 375 mg/day
* No concurrent hormone replacement therapy, tamoxifen, or raloxifene
* Concurrent oral contraceptives allowed provided the dose has not been changed for at least 6 months prior to study entry
* No concurrent chemotherapy or radiation therapy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose that causes 25% DLT assessed using NCI CTCAE version 3.0 | 6 months

SECONDARY OUTCOMES:
Breast tissue histology (nonproliferative, proliferative without atypia, atypical hyperplasia) | Up to 6 months
  Generalized linear models will be used.
COMT genotype | Up to 6 months
  Generalized linear models will be used.
Quality-of-life measures assessed using SF-36 | Up to 6 months
  Generalized linear models will be used.
Protein expression levels in benign breast tissue (Ki-67, p53, EGFR, HER2/neu, cleaved caspase-3, and ER) | Up to 6 months
  Generalized linear models will be used.
Quantitative mammographic breast density | Up to 6 months
  Generalized linear models will be used.
Hormone metabolite levels (estradiol, testosterone, IGF-1, IGFBP-3, SHBG) | Up to 6 months
  Generalized linear models will be used.
Eicosanoid levels (urine PGE-M) | Up to 6 months
  Generalized linear models will be used.
Levels of oxidative damage biomarkers (urine 8-OHdG, isoprostane) | Up to 6 months
  Generalized linear models will be used.
Serum CRP levels | Up to 6 months
  Generalized linear models will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Crew KD, Brown P, Greenlee H, Bevers TB, Arun B, Hudis C, McArthur HL, Chang J, Rimawi M, Vornik L, Cornelison TL, Wang A, Hibshoosh H, Ahmed A, Terry MB, Santella RM, Lippman SM, Hershman DL. Phase IB randomized, double-blinded, placebo-controlled, dose escalation study of polyphenon E in women with hormone receptor-negative breast cancer. Cancer Prev Res (Phila). 2012 Sep;5(9):1144-54. doi: 10.1158/1940-6207.CAPR-12-0117. Epub 2012 Jul 24. PMID 22827973